CLINICAL TRIAL: NCT01540682
Title: Phase I Study of MLN8237 in Combination With Cetuximab and Definitive Radiation in Patients With Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: MLN8237 in Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 10311
Record Dates: First submitted 2012-02-09; First posted 2012-02-29 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Cancer
Keywords: Male and female patients with HNSCC of the oral cavity, oropharynx, hypopharynx, larynx,; nasopharynx or paranasal sinuses that is considered appropriate; for definitive cetuximab-based radiation therapy.
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases | interventions — MLN 8237; Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MLN8237 — Three dose levels of MLN8237 are planned:30, 40 and 50 mg po bid.
Drug: Cetuximab — ~ 1 week prior to the initiation of radiation therapy and continuing for a grand total of 12 weeks.
Radiation: Radiotherapy — Radiotherapy will be administered in 2-Gy fractions, 5 days a week to a total dose of ~70 Gy.

SUMMARY:
This study will evaluate the initial safety and effectiveness of an investigational drug, MLN8237, added to routine radiation therapy and cetuximab in patients with head and neck cancer. This study will also determine the highest dose of MLN8237 that can be given together with cetuximab and radiation therapy without causing severe side effects.

DETAILED DESCRIPTION:
This is a phase 1b study of MLN8237, cetuximab and definitive radiation therapy for patients with previously untreated locoregionally advanced HNSCC who are candidates for definitive radiation therapy with curative intent with cetuximab as the radiosensitizer. The treatment regimen consists of MLN8237 po bid for 7 days followed by 2 weeks off for 4 cycles with the first 3 cycles of MLN8237 concurrent with RT. Three dose levels of MLN8237 are planned: 30, 40 and 50 mg po bid. Cetuximab will be given at the FDA-approved loading and maintenance doses starting ~ 1 week prior to the initiation of radiation therapy and continuing for a grand total of 12 weeks. Radiotherapy will be administered in 2-Gy fractions, 5 days a week, to total dose of ~70 Gy according to standard departmental protocols. Correlative biomarker assays on pre- and on-therapy biopsy specimens (tissue micro arrays analyzed by AQUA quantitative immunofluorescence) will seek to establish proof-of-mechanism by determining if the novel drug combination has the predicted effects on biochemical signaling pathways linked to Aurora A and EGFR. Tumor samples will also be analyzed for Aurora A and EGFR expression by IHC and FISH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females greater than 18 years of age.
2. ECOG performance status of 0-1
3. Patients must have histologically or cytologically confirmed HNSCC of the oral cavity, oropharynx, hypopharynx, larynx, nasopharynx or paranasal sinuses that is considered after a multidisciplinary evaluation (surgery, medical oncology & radiation oncology) to be appropriate for definitive cetuximab-based radiation therapy
4. No distant metastatic disease. Minimum work-up includes:

   * History/physical examination within 4 weeks prior to registration, including assessment of weight and weight loss in past 6 months and an examination by a Medical Oncologist
   * PET/CT scan within 6 weeks prior to registration
   * CT scan or MRI of the head and neck (of the primary tumor and neck nodes) within 4 weeks prior to registration
5. Adequate organ and marrow function
6. Negative pregnancy test within 2 weeks prior to registration for women of childbearing potential. The effects of MLN8237 on the developing human fetus are unknown. For this reason and because MLN8237 agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
7. Male subject agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of MLN8237.
8. Ability to understand and willingness to sign a written informed consent document with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Systemic anti-neoplastic treatment within 21 days preceding the first dose of MLN8237. Patients treated with non-cytotoxic small molecule drugs (eg, tyrosine kinase inhibitors, such as erlotinib and hormonal agents, such as letrozole) must not have received treatment with these drugs for at least 2 weeks before the first dose of MLN8237 is administered.
2. Patient has already had definitive surgical treatment, excluding diagnostic biopsy of the primary site or nodal sampling of neck disease. Prior radical or modified neck dissection is also not permitted.
3. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
4. Primary tumor site is skin or salivary gland.
5. Uncorrected CTCAE, v. 4.0 grade 3-4 electrolyte abnormalities
6. Patients may not be receiving any other investigational agents or treatment with any investigational products within 21 days before the first dose of study drug.
7. Patients with known brain metastasis are excluded from this clinical trial because of their poor prognosis and because they often develop rapid progressive neurologic dysfunction that would confound the evaluation of neurological and other adverse events.
8. History of known allergic reactions attributed to compounds of similar chemical or biologic composition to MLN8237 or cetuximab.
9. Patients may not be taking proton pump inhibitors, H2 antagonists or pancreatic enzyme replacement. Subjects who refuse to limit use of alcohol are also excluded.
10. Severe, active co-morbidity
11. Clinical evidence of intestinal malabsorption. Examples include resection of pancreas or upper small bowel, requirement for pancreatic enzymes, or any other condition that would modify small bowel absorption of oral medications.
12. Prior treatment with high-dose chemotherapy, defined as chemotherapy requiring the use of peripheral blood or bone marrow stem cell support for hematopoietic reconstitution, including prior allogeneic bone marrow transplantation.
13. Prior radiotherapy to greater or equal to 25% of bone marrow. Whole pelvic radiation is considered to be over 25%.
14. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
15. Major surgery within 14 days prior to the first dose of study drug treatment.
16. Inability to swallow oral medication or to maintain a fast as required 2 hours before and 1 hour after MLN8237 administration.
17. Known history of HIV infection, or active hepatitis B, or hepatitis C infection. Testing is NOT required in the absence of clinical findings or suspicion.
18. Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen.
19. Patient has Grade 2 or higher peripheral neuropathy within 14 days before enrollment.
20. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum -human chorionic gonadotropin (-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
21. Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Roger Cohen, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States